CLINICAL TRIAL: NCT03451188
Title: Impact Study on Cerecare Compression Garments in the Treatment of Ehlers-Danlos Syndromes
Status: Completed | Type: Observational
Sponsor: Cerecare (Industry)
Responsible Party: Sponsor
Other Study IDs: SEDCARE
Record Dates: First submitted 2018-01-23; First posted 2018-03-01 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: Eds, Unspecified Type
MeSH Terms: conditions — Ehlers-Danlos Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Cerecare compression garments — all Cerecare compression garments

SUMMARY:
EDS (Ehlers-Danlos syndromes) form a heterogeneous group of hereditary connective tissue pathologies, which present a characteristic triad: cutaneous hyperelasticity, articular hyperlaxity and connective tissue fragility.

The innumerable sprains and dislocations of all the joints require recurrent immobilizations and are responsible for a musculoskeletal handicap, chronic pains and a great fatigability, resounding on the quality of life of the patient.

The use of custom-made compression garments seems to provide relief from pain, especially nociceptive pain and in stabilizing joints by proprioceptive effect.

The SEDCARE study is an observational monocentric, non-comparative study. 76 patients will be followed in this study for 2 years during which they will wear compression custom-made garments (Cerecare®).The main objective of this study is to demonstrate the effectiveness of pressure garments Cerecare in the EDS, especially in terms of joint pain.

ELIGIBILITY:
Inclusion Criteria:

* Ehlers-Danlos syndrome diagnosis confirmed by a medical specialist, according to the new diagnostic criteria of 2017,
* Articular hyperlaxity,
* Have not used compression garments for at least 1 year,
* Without expected body weight change within 6 months,
* Having agreed to participate in the study

Exclusion Criteria:

* Presenting a known allergy to the components of compression garments,
* Presenting acute and unusual pain, not medically controlled,
* Pregnant woman,
* Participating simultaneously with another study or having recently participated in another study for which the exclusion period would not be completed.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: EDS patient
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Joint pain assessment | 6 months
  Assessment of the most painful joint by an VAS (Visual Analog Scale) [0-100mm]. The most painful joint at 0 months (= before use Compression Garments) will be choose as the primary outcome measure. The primary outcome measure will be done at 6 months.

SECONDARY OUTCOMES:
Joint pain assessment | 6, 12, 18 and 24 months
  Assessment of joint pain by an VAS (Visual Analog Scale) [0-100mm]: shoulder, elbow, wrist, finger, hip, knee, ankle.
Daily monitoring of joint instability | 6, 12, 18 and 24 months
  Daily monitoring of joint instability as sprain, dislocation and subluxation (shoulder, elbow, wrist, finger, hip, knee, ankle).
Neuropathic pain assessment | 6, 12, 18 and 24 months
  Assessment of neuropathic pain by the PAIN Detect questionnaire.
  The PAIN Detect questionnaire contains:
  * 3 numerical scales (NS) [0-10],
  * 7 items with categorical response (never, hardly noticed, slightly, moderately, strongly, very strongly).
Proprioception disorders | 6, 12, 18 and 24 months
  Assessment of proprioception disorders by the Berg Balance Scale (BBS) [0-56]. The BBS contains 14 items; each item is scored from 0 to 4.
Functional independence assessment | 6, 12, 18 and 24 months
  Assessment of functional independence by the Functional Independence Measure (FIM) [18-126].
  The FIM contains 18 items; each item is scored from 1 (total assistance) to 7 (complete independence).
Tiredness | 6, 12, 18 and 24 months
  Assessment of Tiredness by the FSS scale (Fatigue Severity Scale) [1-7].
Patient's quality of life | 6, 12, 18 and 24 months
  Assessment of Life quality by the SF-12 questionnaire (Short Form questionnaire on quality of life with 12 items).
Tolerance: incidence of Treatment-Emergent Adverse Events | 6, 12, 18 and 24 months
  By questioning the patient and by a medical exam, evaluation of adverse effect due to compression garments (Yes/ No): itch, edema, blister, redness, dermal ulceration.
Compliance | 6, 12, 18 and 24 months
  By questioning the patient, estimate the number of hours of compression garments daily use.

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Dr Pontier, Clermont-Ferrand
  - Dr Benistan, Garches
  - Dr Michot, Paris
  - Dr Enjalbert, Perpignan
  - SLB Pharma, Rennes